CLINICAL TRIAL: NCT00693667
Title: A Phase II, Double-Blind, Randomized, Placebo-controlled, Clinical Study of PH3 for the Prevention of Osteoporosis in Postmenopausal Women
Brief Title: Study of PH3 for the Prevention of Osteoporosis in Postmenopausal Women
Acronym: PH3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PhytoHealth Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PH-CP011; 93-EC-17-A-17-I1-0034
Record Dates: First submitted 2008-02-19; First posted 2008-06-09 (Estimated); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Osteoporosis
Keywords: osteoporosis; postmenopausal women; botanical drug
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Placebo Comparator): Placebo
  Interventions: Drug: PH3
- B (Active Comparator): 250 mg active ingredient
  Interventions: Drug: PH3
- C (Active Comparator): 500 mg active ingredient
  Interventions: Drug: PH3
- D (Active Comparator): 750 mg active ingredient
  Interventions: Drug: PH3

INTERVENTIONS:
Drug: PH3 — Each PH3 tablet, 530 mg/tablet, contains 250 mg of active ingredient. The placebo tablet contains no active ingredient. Three tablets per day will be taken orally before bedtime.

SUMMARY:
The primary objective of this clinical study is to evaluate the effectiveness and safety of PH3 for the prevention of osteoporosis.

The secondary objectives are to identify the optimal dosage for subsequent studies and to provide basis for the next confirmatory study in study design, endpoints, and study methodologies.

ELIGIBILITY:
Inclusion Criteria:

1. Women 40-60 years of age.
2. Must be postmenopausal (0.5~5 years post cessation of menses) or ovariectomized or hysterectomy women who have documented elevated Follicle Stimulating Hormone FSH (>30mIU/ml) with low serum estradiol (<20 pg/ml).
3. The lumbar vertebral BMD T-score is between -1and -2.5 SD.
4. The body mass index (BMI) is between 19 and 29 kg/m2.
5. Completed informed consent and signed informed consent form.

Exclusion Criteria:

1. Have diseases which may affect bone metabolism, e. g., hyper-or hypocalcemia, hyperthyroidism, osteogenesis imperfecta, malignancy, chronic gastrointestinal disease, extensive Paget's disease, alcoholism, and renal or hepatic impairment.
2. Has taken drug therapy for osteoporosis within the previous six months (excluding calcium supplements) prior to this study.
3. Chronic or continued use of hormone replacement drugs or medications that may affect bone calcium metabolism, for example, phosphate-binding antacids, many diuretics, adrenal or anabolic steroids, heparin, anticonvulsants, fluoride in excess of 1 mg/day and supplements of vitamin D or A in excess of RDAs.
4. Vitamin D deficiency (1, 25-dihydroxyvitamin D is lower than the normal range of: 25.1 pg/mL ~ 66.1 pg/mL).
5. Patients with fracture history.
6. Patients who can not promise to keep from taking stimulant drinks (for example, coffee, tea, alcoholic drink, and Coke) that may cause loss of bone calcium, during the study period.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2008-02; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Biochemical Markers | four weeks

SECONDARY OUTCOMES:
Bone Densitometry | four weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hsiang Tai Chao, Ph.D, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veteran General Hospital, Taipei, Taiwan